CLINICAL TRIAL: NCT05265091
Title: An Open, Multi-Center Phase I/II Clinical Study To Evaluate The Safety, Tolerability, Pharmacokinetic Characteristics And Effectiveness Of KL590586 Capsules In Patients With Advanced Solid Tumors Carrying RET Fusion Or Mutant Genes
Brief Title: A Study of KL590586 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL400-Ⅰ/Ⅱ-01
Record Dates: First submitted 2022-02-14; First posted 2022-03-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
Keywords: Lung; NSCLC; Thyroid
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KL590586 (Experimental): Multiple doses of KL590586 capsule
  Interventions: Drug: KL590586 Capsule

INTERVENTIONS:
Drug: KL590586 Capsule — Product Name: KL590586 Capsules Formulation：Capsule Specification: 10mg; 50mg Ingredients: KL590586, microcrystalline cellulose, mannitol, cross-linked sodium carboxymethylcellulose, colloidal silicon dioxide, magnesium stearate, hydroxypropylmethylcellulose hollow capsule

SUMMARY:
An Open, Multi-Center Phase I/II Clinical Study To Evaluate The Safety, Tolerability, Pharmacokinetic Characteristics And Effectiveness Of KL590586 Capsules In Patients With Advanced Solid Tumors Carrying RET Fusion Or Mutant Genes

DETAILED DESCRIPTION:
This is an open, multicentre phase I/II study. To evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic properties and efficacy of KL590586 in patients with advanced NSCLC, MTC and other solid tumours carrying a RET fusion or mutation gene. Phase I of this study includes a dose-escalation phase and a dose-expansion phase (as needed), which will focus on exploring MTD and/or RP2D of KL590586 in patients with advanced solid tumours; Phase II will assess the efficacy and safety of KL590586 in different cohorts (NSCLC, MTC and other tumour types carrying RET fusions or mutations) of solid tumour patients at the RP2D dose.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I: locally advanced or metastatic solid tumors that are pathologically diagnosed without standard treatment or intolerant to standard treatments
2. Stage II: locally advanced or metastatic NSCLC, MTC or other solid tumors confirmed by pathology
3. There is at least one measurable target lesion that meets RECIST v1.1 or RANO (only for brain tumor lesions)
4. Age > or = 18 years old at the time of signing the informed consent form, regardless of gender
5. Within 14 days before the first administration of the study treatment, the Eastern Cooperative Oncology Group (ECOG) performance status score was 0 or 1, and there was no sudden deterioration, and the expected survival time was > or = 3 months
6. Sufficient organ and bone marrow function (without receiving blood transfusion, erythropoietin, recombinant human thrombopoietin or colony stimulating factor therapy, renal replacement therapy, etc. within 7 days before the examination, the laboratory examination meets the following conditions Regulations): a) Blood routine: absolute neutrophil count (ANC) > or = 1.0×10^9/L; platelet count (PLT) > or = 75×10^9/L; hemoglobin concentration > or = 9.0 g/dl; b) Liver function: AST and ALT < or = 2.5×upper limit of normal (ULN), TBIL< or = 1.5×ULN; for patients with liver metastasis or primary biliary tract tumors, ALT and AST < or = 5×ULN; for liver cancer, liver metastasis or Gil Patients with Gilbert's syndrome, TBIL < or = 3×ULN; c) Renal function: serum creatinine (Cr) < or = 1.5×ULN or creatinine clearance > or = 40 ml/min (using the standard Cockcroft-Gault formula); d) Coagulation function: International normalized ratio (INR), activated partial thromboplastin time (APTT) and prothrombin time (PT) < or = 1.5×ULN;
7. Able to understand and voluntarily sign an informed consent form, and be able to comply with the visit and related procedures stipulated in the plan

Exclusion Criteria:

1. There are known major driver gene changes other than RET. For example, NSCLC carrying targeted mutations such as EGFR, ALK, ROS1 or BRAF; colorectal cancer carrying mutations such as oncogenic KRAS, NRAS or BRAF. If the patient has a co-mutation, the investigator should discuss with the sponsor whether the patient can be included in the group
2. Symptomatic primary central nervous system (CNS) tumors, brain metastases, leptomeningeal carcinogenesis, or untreated spinal cord compression that the researchers believe require local intervention
3. People with other active malignant tumors (except for non-melanoma skin cancer in situ, cervical cancer in situ and other localized tumors that have been cured and have not recurred within 5 years)
4. Need to use drugs known to be potent inhibitors or inducers of CYP3A4, drugs known to prolong QTc, and the treatment cannot be terminated at least 14 days before the study drug is administered
5. Received the following anti-tumor treatments: a) The previous anti-tumor drug treatment (except immunotherapy or other antibody therapy) is less than 14 days or 5 half-lives (whichever is longer) from the first treatment with study drug; b) In Those who have received any immunotherapy or other antibody treatment within 28 days before the first study drug administration; c) Those who have received more than 30% of bone marrow radiation or wide-range radiotherapy within 28 days before the first study drug treatment (the patients receiving palliative radiotherapy are the first Within 7 days before receiving study drug treatment)
6. Received major surgical operations within 28 days before receiving the first study drug treatment (excluding operations such as central venous catheter placement, tumor biopsy, and gastric tube placement)
7. Those who have received other clinical trial drug treatment within 28 days before receiving the first study drug treatment
8. Any original symptoms that may interfere with the results of the study, including: any unrecovered toxicity above grade 1 of the CTCAE related to previous anti-tumor therapy (hair loss and grade 2 neuropathy related to previous platinum-based drug treatment, etc.) Except for chronic toxicity judged by the person
9. Patients with clinically active interstitial lung disease, active pneumonia, and radiation pneumonia requiring treatment, or those who have been found or suspected of having such diseases during the screening period
10. Poorly controlled pleural effusion, abdominal effusion, or pericardial effusion after intervention (such as drainage)
11. Any serious and/or uncontrolled comorbidities that may prevent the patient from participating in the study
12. Those who are known to be allergic to any component in the study drug prescription
13. Clinically significant active malabsorption syndrome or other diseases that may affect study drug administration and gastrointestinal absorption
14. Active hepatitis B (hepatitis B surface antigen is positive and HBV-DNA is higher than the upper limit of normal detection) or hepatitis C (hepatitis C antibody is positive and HCV-RNA is higher than the upper limit of normal detection); Human immunodeficiency virus (HIV) examination Positive or known acquired immunodeficiency syndrome (AIDS); Treponema pallidum antibody test is positive
15. Pregnant or breastfeeding women, fertility patients (regardless of male and female) who cannot take effective medical contraceptive measures during the study period and within 6 months after the last administration
16. Other situations where the researcher thinks it is inappropriate to participate in this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose limiting toxicities (DLT) | From date of initial dose until up to 28 days for treatment
  Incidence rate of dose limiting toxicities (DLT)
Phase II: ORR | Approximately 12 months
  Objective response rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Xiangqian Zheng, Professor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Shanghua Jing, Professor, Principal Investigator — The Fourth Hospital of Hebei Medical University and Hebei Cancer Hospital; Anwen Liu, Professor, Principal Investigator — Second Affiliated Hospital of Nanchang University; Yilong Wu, Professor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Sichuan Kelun Botai Biopharmaceutical Co., Chengdu, Sichuan, China